CLINICAL TRIAL: NCT04581239
Title: Effect of Active Versus Passive Lower Extremity Neural Mobilization Combined With Lumbar Traction and Lumbar Mobilization in Patients With Lumbar Radiculopathy
Brief Title: Effect of Active Versus Passive Lower Extremity Neural Mobilization in Lumber Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/19/2025 Hafiz Abdul Rehman
Record Dates: First submitted 2020-10-03; First posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Lumbar Radiculopathy
Keywords: Active Neural Mobilization; Lumber Traction; Lumber Mobilization; Passive Neural Mobilization; Lumber Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active neural mobilization (Active Comparator): Therapist supervised active neural mobilization of sciatic nerve in lumber radiculopathy patients
  Interventions: Other: Active neural mobilization
- passive neural mobilization (Experimental): Therapist done passicive neural mobilization of sciatic nerve in lumber radiculopathy patients
  Interventions: Other: passive neural mobilization

INTERVENTIONS:
Other: Active neural mobilization — Active neural mobilization Base line treatment followed heating pad 10 minutes, lumber traction with 50 %of body weight in accordance with tolerance. 15 to 20 Lumber segmental mobilization.
  Active oscillatory nerve mobilization was given in 3 sets of 10 repetition in each set with 20 sec rest time between set
  Arms: Active neural mobilization
Other: passive neural mobilization — Base line treatment followed heating pad 10 minutes, lumber traction with 50 %of body weight in accordance with tolerance. 15 to 20 Lumber segmental mobilization
  Passive neural mobilization This oscillatory nerve mobilization was given in 3 sets of 10 repetition in each set with 20 sec rest time between set. Both groups received total 18 session 3 session per week for consecutive 6 weeks
  Arms: passive neural mobilization

SUMMARY:
The aim of this study was to find out the effects of active versus passive lower extremity neuralmobilizations combined with lumbar traction and lumbar mobilization in patients with lumbarradiculopathy. The study was conducted in shalamar hospital Lahore and was completed within 6 month of time duration. Sample size of twenty four patient consists of both male and female aged between 45 years to 65 years. Each group contain 12 patients. Group A received active neural mobilizations whereas group B received passive neural mobilization along with lumber traction and mobilization. Patients were re assessed at the end of 6 weeks through SLR , NPRS and ODI.

DETAILED DESCRIPTION:
Lower back pain is found to be one of the common health condition approximately 80% of individual experience back pain once in their lives. Radicular lower back pain is also a disorder that involves the dysfunction of the nerve roots of lumbosacral region. Its symptoms include radiating pain with numbness, paraesthesia and muscle weakness. In general population the annual prevalence of lumber radiculopathy varied from 9.9% to 25% .. Many of the spinal structures notably ligaments, paravertebral muscles, facet joints, spinal nerve roots and annulus fibrosis have been considered as the main cause of the pain. Clinical examinations mostly aim to clarify that whether a nerve root has mechanical impingement. The common clinical diagnostic tests include tests for tendon reflexes, straight leg raise test(SLR), sensory deficits and motor weakness. Several clinicians and researchers have come up with several debates for the treatment of Lower back pain. But not many studies have come up that actually authenticates that how much effective are physical therapy interventions. The common treatments for radical lower back pain includes physical modalities like TENS, ultrasound, Heat and Cryotherapy, lumbar traction and lumbar spinal mobilizations. Kinesiotherapy including ROM exercises and strengthening are also used to treat lower back pain. Neural mobilization techniques actually help in restoring the plasticity of nervous system. Plasticity of nervous system is actually the ability of the nerve surrounding structures to adapt of shift according to other structures. The aim of mobilization is actually to increase the collagen flexibility that helps in maintaining the integrity and movement of the nerve according to its surrounding structures. Radiculopathy management and lower back pain management have a direct link with neural mobilization.

However, evidence lacks whether active or passive lower extremity neural mobilization is more effective. Thus, the purpose of the current study is to compare the effects of active and passive neural mobilization in the management of lumbar radiculopathy, in combination with mechanical traction and joint mobilization.

In 2016 an RCT was conducted and concluded the efficacy of neural mobilization techniques in patients with radicular low back pain. They concluded that neural mobilizations techniques in radicular low back pain are effective. They stated that these techniques reduce the pain, functional disability and enhance the physiological functioning of the nerve root in patients in low back pain with lumbosacral radiculopathy . In 2014 A comparative study was conducted and found that lower extremity neural mobilizations along with conventional physiotherapy such as lumbar traction and lumbar mobilizations improves the agility in lower extremity and reduces pain and disability.

2013 a Study was conducted to observe observed the effects of neural mobilizations in the patients with radicular low back pain and concluded that patients treated with neural mobilizations showed better VAS score. They stated that further research is needed in order to assess the long-term effects of treatment and treatments provided on more than one occasion.

The purpose of the study was to determine the effects of active verses passive lower extremity neural mobilizations combined lumbar traction and lumbar mobilization so that in future this study should be helpful for other researchers to determine which therapy is most helpful in rehabilitation of the patients with radicular low back pain signs and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Pain radiate from lower lumber area to posterior aspect of leg up to planter surface of toes.
* Patient with confirmed L4-L5, L5-S1 disc herniation or disc bulge diagnosed by neurophysician.
* Numeric pain rating scale value is more than 4.
* Patients having positive compression distraction, Lasegue's sign and lower limb neural tension tests. (LLNTT).Lasègue's sign is said to be positive if the angle to which the leg can be raised (upon straight leg raising) before eliciting pain is <45°.

Exclusion Criteria:

* Any red flags (tumor, fracture, metabolic diseases, rheumatoid arthritis, osteoporosis, resting
* blood pressure greater than 140/90 mmHg, prolonged history of steroid use, etc)
* Any systemic disease as diabetes or neurological condition that altered the function of the nervous system
* Prolong use of steroids.
* History of any surgery, trauma, or pathology of back, hip, knee, and ankle.
* Spinal stenosis, Potts disease
* Taking any treatment or medication except physiotherapy

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 6 week
  Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain.

SECONDARY OUTCOMES:
Straight Leg Raise (SLR) | 6 week
  A positive straight leg raising test (also known as Lasegue sign) results from gluteal or leg pain by passive straight leg flexion with the knee in extension, and it may correlate with nerve root irritation and possible entrapment with decreased nerve excursion
Oswestry Disability Index (ODI) questionnaire | 6 week
  The Oswestry Disability Index (ODI)7,9 is the most commonly used outcome-measure questionnaire for low back pain in a hospital setting. It is a self-administered questionnaire divided into ten sections designed to assess limitations of various activities of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, Phd*, Principal Investigator — Riphah International University
Locations (1):
- Shalamar hospital Lahore, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Masters S, Lind R. Musculoskeletal pain - presentations to general practice. Aust Fam Physician. 2010 Jun;39(6):425-8. PMID 20628683
- [Background] Satpute K, Hall T, Bisen R, Lokhande P. The Effect of Spinal Mobilization With Leg Movement in Patients With Lumbar Radiculopathy-A Double-Blind Randomized Controlled Trial. Arch Phys Med Rehabil. 2019 May;100(5):828-836. doi: 10.1016/j.apmr.2018.11.004. Epub 2018 Dec 3. PMID 30521781
- [Background] Ellis RF, Hing WA. Neural mobilization: a systematic review of randomized controlled trials with an analysis of therapeutic efficacy. J Man Manip Ther. 2008;16(1):8-22. doi: 10.1179/106698108790818594. PMID 19119380
- [Background] Hahne AJ, Ford JJ, McMeeken JM. Conservative management of lumbar disc herniation with associated radiculopathy: a systematic review. Spine (Phila Pa 1976). 2010 May 15;35(11):E488-504. doi: 10.1097/BRS.0b013e3181cc3f56. PMID 20421859
- [Background] Harte AA, Baxter GD, Gracey JH. The effectiveness of motorised lumbar traction in the management of LBP with lumbo sacral nerve root involvement: a feasibility study. BMC Musculoskelet Disord. 2007 Nov 29;8:118. doi: 10.1186/1471-2474-8-118. PMID 18047650
- [Background] Boyles R, Toy P, Mellon J Jr, Hayes M, Hammer B. Effectiveness of manual physical therapy in the treatment of cervical radiculopathy: a systematic review. J Man Manip Ther. 2011 Aug;19(3):135-42. doi: 10.1179/2042618611Y.0000000011. PMID 22851876
- [Background] Efstathiou MA, Stefanakis M, Savva C, Giakas G. Effectiveness of neural mobilization in patients with spinal radiculopathy: a critical review. J Bodyw Mov Ther. 2015 Apr;19(2):205-12. doi: 10.1016/j.jbmt.2014.08.006. Epub 2014 Aug 17. PMID 25892373
- [Background] Kawakami M, Weinstein JN, Spratt KF, Chatani K, Traub RJ, Meller ST, Gebhart GF. Experimental lumbar radiculopathy. Immunohistochemical and quantitative demonstrations of pain induced by lumbar nerve root irritation of the rat. Spine (Phila Pa 1976). 1994 Aug 15;19(16):1780-94. doi: 10.1097/00007632-199408150-00001. PMID 7526474
- [Background] Kostadinovic S, Milovanovic N, Jovanovic J, Tomasevic-Todorovic S. Efficacy of the lumbar stabilization and thoracic mobilization exercise program on pain intensity and functional disability reduction in chronic low back pain patients with lumbar radiculopathy: A randomized controlled trial. J Back Musculoskelet Rehabil. 2020;33(6):897-907. doi: 10.3233/BMR-201843. PMID 32675390
- [Background] Winkelstein BA, DeLeo JA. Nerve root injury severity differentially modulates spinal glial activation in a rat lumbar radiculopathy model: considerations for persistent pain. Brain Res. 2002 Nov 29;956(2):294-301. doi: 10.1016/s0006-8993(02)03560-6. PMID 12445698
- [Background] Kobayashi S, Kokubo Y, Uchida K, Yayama T, Takeno K, Negoro K, Nakajima H, Baba H, Yoshizawa H. Effect of lumbar nerve root compression on primary sensory neurons and their central branches: changes in the nociceptive neuropeptides substance P and somatostatin. Spine (Phila Pa 1976). 2005 Feb 1;30(3):276-82. doi: 10.1097/01.brs.0000152377.72468.f4. PMID 15682006
- [Background] Leininger B, Bronfort G, Evans R, Reiter T. Spinal manipulation or mobilization for radiculopathy: a systematic review. Phys Med Rehabil Clin N Am. 2011 Feb;22(1):105-25. doi: 10.1016/j.pmr.2010.11.002. Epub 2010 Dec 30. PMID 21292148
- [Background] Plaza-Manzano G, Cancela-Cilleruelo I, Fernandez-de-Las-Penas C, Cleland JA, Arias-Buria JL, Thoomes-de-Graaf M, Ortega-Santiago R. Effects of Adding a Neurodynamic Mobilization to Motor Control Training in Patients With Lumbar Radiculopathy Due to Disc Herniation: A Randomized Clinical Trial. Am J Phys Med Rehabil. 2020 Feb;99(2):124-132. doi: 10.1097/PHM.0000000000001295. PMID 31464753
- [Background] Han L, Zhao P, Guo W, Wei J, Wang F, Fan Y, Li Y, Min Y. Short-term study on risk-benefit outcomes of two spinal manipulative therapies in the treatment of acute radiculopathy caused by lumbar disc herniation: study protocol for a randomized controlled trial. Trials. 2015 Mar 27;16:122. doi: 10.1186/s13063-015-0634-0. PMID 25872929